CLINICAL TRIAL: NCT01413893
Title: An Extension Study of Linifanib in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: An Extension Study of Linifanib (ABT-869) in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M12-749
Record Dates: First submitted 2011-06-23; First posted 2011-08-10 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-06

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- linifanib (Experimental)
  Interventions: Drug: linifanib

INTERVENTIONS:
Drug: linifanib — QD daily
  Other Names: ABT-869

SUMMARY:
An extension study of linifanib in subjects with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety of linifanib in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria

1. Subject has completed a previous study utilizing linifanib (per the criteria in the previous study) or was active and assigned to linifanib when the study was completed and the investigator believes that continued treatment with linifanib is in the best interest of the subject.
2. Women of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 90 days following completion of therapy. Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential:

   * total abstinence from sexual intercourse (minimum one complete menstrual cycle);
   * vasectomized partner(s);
   * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration; if the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after study completion;
   * intrauterine device (IUD);
   * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or creams);
   * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completion of therapy.
3. Is capable of understanding and complying with parameters as outlined in the protocol and able to sign the informed consent, approved by an Independent Ethic Committee (IEC)/Institutional Review Board (IRB) prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria

1. Subject discontinued linifanib administration before completing the prior study (due to disease progression, toxicity, withdrawal of consent, other).
2. Subject has any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
3. Subject is a lactating or pregnant female.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events - The number of participants with adverse events will be reported as a measure of Safety. | All adverse events occuring through the Final Visit will be reported.
  The investigators will monitor each subject for clinical and lab evidence of adverse events on a routine basis through out the study. The investigators will question each subject regarding any adverse effects that they have experienced and record any events on the care report forms. All adverse events will be followed to a satisfactory clinical resolution.
Safety: Physical Examination and Vital Signs - Physical examination will be performed and vital signs will be assessed for participants as a measure of safety. | Change from baseline to Day 1 of Weeks 1, 2, 3, 6, 9 and 12 and on Week 24 then Day 1 of every 12 weeks and Final Visit.
  Physical exam, blood pressure, pulse, body temperature will be measured and recorded on the case report forms.
Safety: Multiple Gated Acquisition (MUGA) will be assessed at specified time points as a measure of safety. | Change from baseline to every 12 weeks
  MUGA
Safety: Clinical Lab Tests will be performed for each participant as a safety measure. | Change from baseline to Day 1 of Weeks 1, 2, 3, 6, 9 and 12 and on Week 24 then Day 1 of every 12 weeks and Final Visit
  Chemistry, hematology, urinalysis lab tests will be measured and recorded on the case report forms. All clinically significant values will be followed by the investigator to a satisfactory clinical resolution.

SECONDARY OUTCOMES:
There are no secondary outcome measures specified for this study. | There are no secondary outcome measures specified for this study.
  There are no secondary outcome measures specified for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. McKee, MD, Study Director — Abbott